CLINICAL TRIAL: NCT01962376
Title: Phase IV Multi-Institutional Randomized Trial of Capecitabine Plus Oxaliplatin With Bevacizumab in Patients With Potentially Resectable Gastric Cancer With Liver Metastasis
Brief Title: Preoperative Chemotherapy With Bevacizumab For Potentially Resectable Gastric Cancer With Liver Metastasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yan Zhang, The first hospital of Shijiazhuang city, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YZHANG0001
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Cancer; Liver Metastasis
Keywords: Capecitabine; Oxaliplatin; Bevacizumab; Potentially Resectable Gastric Cancer Liver Metastasis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab,postoperative chemotherapy (Active Comparator): Groups 1 drug: Oxaliplatin;Capecitabine;Bevacizumab A cycle:Capecitabine 2000mg/m2 D1-D14 q3wk、Oxaliplatin 130 mg/m2 D1 q3wk add and subtract. Bevacizumab 7.5mg/kg D1 q3wk.Evaluation for every two cycles.
  Groups 2 drug: Oxaliplatin;Capecitabine A cycle:Capecitabine 2000mg/m2 D1-D14 q3wk、Oxaliplatin 130 mg/m2 D1 q3wk.Evaluation for every two cycles.
  placebo:Physiological saline
  Interventions: Drug: Oxaliplatin;Capecitabine; Drug: Oxaliplatin;Capecitabine;Bevacizumab
- Preoperative Chemotherapy (Experimental): Groups 1 drug: Oxaliplatin;Capecitabine;Bevacizumab A cycle:Capecitabine 2000mg/m2 D1-D14 q3wk、Oxaliplatin 130 mg/m2 D1 q3wk add and subtract. Bevacizumab 7.5mg/kg D1 q3wk.Evaluation for every two cycles.
  Groups 2 drug: Oxaliplatin;Capecitabine A cycle:Capecitabine 2000mg/m2 D1-D14 q3wk、Oxaliplatin 130 mg/m2 D1 q3wk.Evaluation for every two cycles.placebo:Physiological saline
  Interventions: Drug: Oxaliplatin;Capecitabine; Drug: Oxaliplatin;Capecitabine;Bevacizumab

INTERVENTIONS:
Drug: Oxaliplatin;Capecitabine — A cycle:Capecitabine 2000mg/m2 D1-D14 q3wk、Oxaliplatin 130 mg/m2 D1 q3wk.Evaluation for every two cycles.
  Other Names: Oxaliplatin plus capecitabine other names:XELOX.
Drug: Oxaliplatin;Capecitabine;Bevacizumab — A cycle:Capecitabine 2000mg/m2 D1-D14 q3wk、Oxaliplatin 130 mg/m2 D1 q3wk add and subtract. Bevacizumab 7.5mg/kg D1 q3wk.Evaluation for every two cycles.
  Other Names: Capecitabine Plus Oxaliplatin Other names XELOX.

SUMMARY:
The investigators assessed whether the addition of a preoperative regimen of Bevacizumab regimen to improves R0 resection rate and survival among patients with potentially resectable gastric cancer with liver metastasis.

DETAILED DESCRIPTION:
Groups 1:Capecitabine Plus Oxaliplatin With Bevacizumab in Patients With Potentially Resectable Gastric Cancer With Liver Metastasis.

Groups 2:Capecitabine Plus Oxaliplatin With placebo in Patients With Potentially Resectable Gastric Cancer With Liver Metastasis.

Group 1 compare with Group 2 in disease-free survival time. Stage I：Preoperative therapy Capecitabine Plus Oxaliplatin With Bevacizumab is superior to Capecitabine Plus Oxaliplatin alines.

Stage II: therapy after surgery Capecitabine Plus Oxaliplatin With Bevacizumab is superior to Capecitabine Plus Oxaliplatin alones after surgery for over 6 months in all.

ELIGIBILITY:
Inclusion Criteria:

* 1.Pathological tissue were gastric cancer by gastric and liver biopsy.

  2.Immunohistochemistry confirmed HER-2 ( - ).

  3.The number of liver metastasis is less than 3 and evey one is less than 5 cm.

  4.Liver metastasis must be clinically limited to Type H1 or Type H2.

  5.gastric cancer were able to resectable lesions or T1-4a N1-2 M0.

  6.Patients•had not received radiotherapy past and not other organ metastasis and peritoneal metastasis.

  7.Karnofsky performance status performance status >70.

  8.Inadequate hematopoietic function： Hemoglobin≥90g/L; ANC≥1,500/mm3;Platelet≥100,000/mm3

  9.Inadequate organ function which is defined as below: Total bilirubin≤1.5 pper limit of normal range (ULN);alanine transaminase / Aspertate aminotransferase≤2.5 upper limit of normal range (ULN) (≤5.0 x ULN if hepatic metastasis); serum creatinine≤1.5 pper limit of normal range (ULN), Serum albumin≥30g/L.

  10.expectancy must be more than 3 months.

  11.the random blood or urine pregnancy test in fertile woman must be the negative results in pregnancy test in 7 days.

  12.Patients for male and female used reliable contraception contraceptive method until the end of study 30 days later.

Type H1: only one leaf with liver metastasis. Type H2: two leaves with a few scattered metastatic in liver.

Exclusion Criteria:

* 1. Patients with other extrahepatic metastasis Include peritoneal metastasis.

  2. Primary was ulcerative type or the existence of the perforation.

  3. Patients with other malignancy in 5 years.

  4. Patients with severe liver disease, kidney disease, respiratory disease , uncontrolled diabetes or severe infections.

  5.Patients with hypertension failed to control, active bleeding, 3~4 proteinuria, heal the wound, thromboembolisms, heart failure, clinical symptoms of heart disease.

  6.Patients have obvious peripheral nervous system disorders,mental disorders and disorders of the central nervous system history.

  7.Patients have history of organ transplantation.

  8.Patients with any medical or psychiatric condition or disease which, in the investigator's judgment, would make the patient inappropriate for entry into this study.

  9.Patients combined antitumor drug outside the research program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | within 3 weeks after surgery

OTHER OUTCOMES:
R0-resection rate | within 3 weeks after surgery
Overall survival (OS) | 2 years
Adverse events | 2 years
  Side effects during observation] Investigators graded all adverse events and toxic effects according to the National Cancer Institute's Common Toxicity Criteria, version 2.0. The number of Participants with adverse events will be recorded at each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, Doctor, Principal Investigator — Hebei Medical University
Locations (1):
- Department of Internal Medicine-Oncology, Shijiazhuang, Hebei, China